CLINICAL TRIAL: NCT06745700
Title: Impact of Behavioral Activation on Depression, Anxiety, Health-related Quality of Life (HRQoL), Cancer Recurrence and Survival in Patients with Colon Cancer
Brief Title: Impact of Behavioral Activation on Depression and Quality of Life in Patients with Colon Cancer
Acronym: BAdepCa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Catarina Tiselius, MD, PhD, Assoc. professor, Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTV-1011976
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Depression - Major Depressive Disorder; Anxiety; Colon Cancer
Keywords: depression; anxiety; health related quality of life; colon cancer
MeSH Terms: conditions — Anxiety Disorders; Colonic Neoplasms; Depression

STUDY DESIGN:
Intervention Model Description: Behavioral: Brief Behavioral Activation
  A five-session telephone-based brief behavioral activation treatment.
  Session 1: Psychoeducation about depression; treatment rationale for Behavioral Activation (BA); rationale and instructions for activity log.
  Session 2: Discussion of life goals and values; planning of activities aligned with life goals and values for coming week.
  Session 3-4: Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for coming week.
  Session 5: Troubleshooting any problems carrying out activities; reviewing treatment; stressing the importance of continuing to engage in activities aligned. with life goals and values; creating a a maintenance plan.
  Other group: care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Behavioural Activation (Experimental): Five-session Brief Behavioral Activation intervention. Sessions 1 - 4 are completed once a week, and session 5 is a booster-session completed four weeks after session 4 and care as usual provided by Region Västmanland.
  Interventions: Behavioral: Brief Behavioural Activation; Other: Care as usual
- Care as Usual (Other): Care as usual provided by Västmanland County hospital.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Brief Behavioural Activation — Behavioral: Brief Behavioral Activation.
  A five-session telephone-based brief behavioral activation treatment.
  Session 1: Psychoeducation about depression; treatment rationale for Behavioral Activation (BA); rationale and instructions for activity log.
  Session 2: Discussion of life goals and values; planning of activities aligned with life goals and values for coming week.
  Session 3-4: Troubleshooting any problems carrying out activities; planning activities aligned with life goals and values for coming week.
  Session 5: Troubleshooting any problems carrying out activities; reviewing treatment; stressing the importance of continuing to engage in activities aligned. with life goals and values; creating a a maintenance plan.
  Other group: care as usual.
  Arms: Brief Behavioural Activation
Other: Care as usual — Care as usual provided by Region Västamanland,

SUMMARY:
The purpose of this randomized clinical trial is to study anxiety and depression symptoms at diagnosis in patients with colon cancer. Previous studies have shown that so-called. Behavioural activation as therapy for these symptoms has a positive impact on the patient's well-being, but it has not been studied whether it also has a positive impact on the patient's mental health in cancer, and whether it can have a prognostically beneficial effect on cancer recurrence risk and survival.

The investigators will investigate the prevalence of anxiety and depression symptoms as well as quality of life in colon cancer patients at diagnosis and at follow-up using self-estimated validated protocols in a prospective cohort study. Data will be compared with data from a reference population. In the cohort study the investigators will also perform a nested randomized clinical trial of a brief psychological treatment called Behavioural Activation to patients with colon cancer and comorbid anxiety and/or depression.

All participants will answer the questionnaires at diagnosis, after1, 2 and 6 months and after 1 and 3 years.

DETAILED DESCRIPTION:
Colon cancer is common. At diagnosis, about 20% have metastatic disease. The prognosis is determined by the stage of the tumour and the degree of spread, but also by the patient's physical health and other diseases. However, it is not known how the patient's mental health are affected and how common anxiety and depression symptoms are at diagnosis. Depression is known to be one of the most common causes of ill health in the world. It also has been shown that patients with depression and cancer also have a poorer survival rate compared to cancer patients without depression However, previous studies have shown that so-called brief Behavioural activation as therapy for these symptoms has a positive impact on the patient's well-being, but it has not been studied whether it also has a positive impact on the patient's mental health in cancer, and whether it can have a prognostically beneficial effect.

The goal of this randomized study is to increase knowledge about, to detect and treat anxiety and depression symptoms in patients with colon cancer, with so-called brief behavioural activation, which can lead to improved care, and possibly improve the patients' prognosis in the form of reduced risk of cancer recurrence and improved survival.

All participants will continue their care as usual (CAU), and half of the participants will be randomized to receive a five-session telephone-based BA-treatment spread over two months as an add-on to CAU. All participants will answer a questionnaire in the beginning of the study, 4 weeks after diagnosis, after 9 weeks, and after 3-, 6- and 12 months.

The main questions that the trial aims to answer are if the BA-treatment has an effect in the short and long term on:

* Depressive symptoms
* Anxiety symptoms
* Self-rated activation
* Self efficacy
* Mental wellbeing
* Quality of life
* Cancer recurrence and survival

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with colon cancer in Region Västmanland, will be considered for inclusion. Those who meet the inclusion criteria will be offered to participate in the studies after written approval.

Exclusion Criteria:

* language difficulties that cause patients to be unable to absorb the treatment
* ongoing alcohol or substance use syndrome
* elevated suicide risk
* ongoing psychotic disorder, severe depression
* antidepressant treatment initiated within the last month
* ongoing or previous manic episode
* cognitive illness/dementia
* ongoing psychological treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Depression Symptoms: Hospital Anxiety and Depression Scale, HADS | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 6 months, 1 and 3 years post-intervention or equivalent for control group.
  The HADS consists of 14 questions, of which 7 constitute a depression scale and 7 constitute an anxiety scale. The points from the seven different statements per subscale are added together and can amount to a maximum of 21 points per subscale. Min 0 and maximum 42 points. Higher scores indicate more anxiety and depression symptoms.
Mental well-being | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 6 months, 1 and 3 years post-intervention or equivalent for control group.
  The short version of the Warwick-Edinburgh Mental Well-being Scale, SWEMWBS. The scores from the seven statements are summed up and vary between minimum 7 and maximum 35 points. Higher scores indicate better psychological well-being.
Health-related quality of life (HRQoL ) | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 6 months, 1 and 3 years post-intervention or equivalent for control group.
  EuroQol-5 Dimensions-5 Level Scale, EQ-5D-5L (Feng et al., 2021). The self-assessment scale consists of sub-questions; five questions with five different answer options where the score varies between 1-5 points, where higher scores indicate better HRQoL.
Behavioral Activation for Depression Scale - Short Form BADS-SF | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 6 months, 1 and 3 years post-intervention or equivalent for control group.
  Rating scale with two subscales where one scale sums up activation and the other about avoidant behavior. The scale varies between 0-54 points, with higher scores indicating more activation.
Perceived self-efficacy | Baseline; post-intervention or equivalent for control group 9 weeks after baseline; 6 months, 1 and 3 years post-intervention or equivalent for control group.
  Swedish translation of The New General Self-Efficacy Scale S- GSE. The total score of the rating scale varies between 10-40 points where higher scores indicate a higher self-perceived self-efficacy.

OTHER OUTCOMES:
Prognostic markers | Measurement 3 and 5 years after diagnosis and treatment.
  Recurrence (3 and 5 years), metastasis (local recurrence and distant metastases), cause of deathe and survival (DFS and OS at 3 and 5 years).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical research and Dept. of Surgery, Västerås, Region Västmanland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified outcome measure IPD will be shared upon reasonable requests from academic researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan to be shared/published before data collection has ended.
Access Criteria: Data will be shared upon reasonable requests assessed by the investigators.

REFERENCES:
- [Background] Pellas J, Renner F, Ji JL, Damberg M. Telephone-based behavioral activation with mental imagery for depression: A pilot randomized clinical trial in isolated older adults during the Covid-19 pandemic. Int J Geriatr Psychiatry. 2022 Jan;37(1):10.1002/gps.5646. doi: 10.1002/gps.5646. Epub 2021 Nov 10. PMID 34729823
- [Background] Funderburk JS, Pigeon WR, Shepardson RL, Maisto SA. Brief behavioral activation intervention for depressive symptoms: Patient satisfaction, acceptability, engagement, and treatment response. Psychol Serv. 2020 Nov;17(4):443-451. doi: 10.1037/ser0000328. Epub 2019 Feb 4. PMID 30714752